CLINICAL TRIAL: NCT06423131
Title: TCRαβ+ Cell Deleted Versus Traditional Haploidentical Hematopoietic Stem Cell Transplantation ：A Single-center, Prospective, Non-randomized Controlled Clinical Study
Brief Title: Prospective Clinical Trial for Children With TCRαβ Depleted vs Traditional Haplo Identicle HSCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sijia Gu (Other)
Responsible Party: Sponsor-Investigator, Sijia Gu, Principal investigator, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCMCIRB-K2024030-2
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Graft-Versus-Host Disease; Hematopoietic Stem Cell Transplantation; Child, Only; Haploidentical Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Intervention Model Description: TCRαβ depleted HSCT compare to traditional Beijing haploidentical HSCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Haplo identicle HCT (No Intervention): Beijing haploidenticla HCT is the routinely traditional way used for haploidentical HCT
- TCRαβ Depleted haploidentical HCT (Experimental): TCRαβ Depleted haploidentical HCT is experimental used to decrease GVHD and obtain better qulity of life for children with haploidentical HCT.
  Interventions: Procedure: TCRαβ Depleted haploidentical HCT

INTERVENTIONS:
Procedure: TCRαβ Depleted haploidentical HCT — Use the CliniMACS TCRα/β deplete from the mobilized peripheral blood stem cells of haploidentical donor in children
  Arms: TCRαβ Depleted haploidentical HCT

SUMMARY:
This is a single-center prospective, non-randomized controlled clinical study in China using CliniMACS TCRα/β+ cell depleted stem cell haploidentical donors versus conventional Beijing protocol for haploidentical hematopoietic stem cell transplantation in children.

DETAILED DESCRIPTION:
1:1 non-randomized controlled clinical study in single center using CliniMACS TCRα/β+ cell depleted stem cell versus conventional Beijing protocol for haploidentical hematopoietic stem cell transplant. The purpose of this study is to obtain 30% decrease grade II-IV aGVHD and better qulity of life for TCRα/β+ cell depleted haploidentical stem cell transplantaion.

ELIGIBILITY:
Inclusion Criteria:

* Age 8 weeks to 18 years
* Children who meet the indicators haploidentical hematopoietic cell transplantation
* No HLA ≥ 9/10 donor or not suitable for this type of donor due to illness
* Informed consent must be signed (by the patient or legal representative)

Exclusion Criteria:

* Liver function abnormalities with bilirubin >2 mg/dL and elevation of transaminases higher than 400 U/L
* Chronic active viral hepatitis
* Ejection fraction <50%
* Respiratory failure necessitating supplemental oxygen
* Patients with a history of psychiatric illness or a condition which could interfere with their ability to understand the requirements of the study
* Patients unwilling or unable to comply with the protocol or unable to give informed consent
* Concurrent severe or uncontrolled infection

Ages: 8 Weeks to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-05-26 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade II-IV acute GVHD | day+100
  Incidence of grade II-IV acute graft-versus-host disease (GVHD) until Day 100 post-transplantation.
incidence of treatment related mortality(TRM) | day +100
  compare the incidence of TRM until Day 100 post-transplantation

SECONDARY OUTCOMES:
post HSCT day 1y and 2y GRFS and OS | day +1y and +2y
  compare the incidence of GRFS and OS post HSCT 1y and 2y
cGVHD post day 1y and 2y | day +1y and +2y
  compare the incidence of cGVHD post HSCT 1y and 2y
TRM post day +1y and +2y | day +1y and +2y
  compre the incidence of TRM post HSCT day 1y and 2y

CONTACTS AND LOCATIONS:
Overall Officials: Jing Chen, PhD, Principal Investigator — Shanghai Children's Medical Center
Locations (1):
- Shanghai Children's Medical Center, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No